CLINICAL TRIAL: NCT01436604
Title: Early Detection of Cardiac Toxicity of Trastuzumab (Herceptin ®) in Patients Treated for Breast Carcinoma: Value of Magnetic Resonance Imaging
Acronym: MRTOX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MRTOX
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Cancer, Breast; LV Dysfunction
Keywords: cardiac MRI; Cancer; Breast; Herceptin; LV dysfunction
MeSH Terms: conditions — Breast Neoplasms; Ventricular Dysfunction, Left; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LV dysfunction group (Other): Cardiac MRI
  Interventions: Other: Cardiac MRI
- Control group (Other): Cardiac MRI
  Interventions: Other: Cardiac MRI

INTERVENTIONS:
Other: Cardiac MRI — The examinations will be conducted on an MRI with a dedicated antenna heart, by a physician with expertise in cardiac MRI.
  After establishing a good quality ECG synchronization, the following sequences are carried out successively:
  * Sequences locating anatomical
  * T2 black blood (such as ESF)
  * rapid sequence of cine-MRI (such as balanced FFE) vertical and horizontal long axis and short axis of the base to the apex
  * T1-weighted sequence with inversion recovery for the assessment of possible consequences of cell damage.

SUMMARY:
The main objective of this study is to compare the proportions of late enhancement in patients with Left ventricular (LV) dysfunction as Herceptin ® and in a control group consisting of patients who did not have LV dysfunction after 6 months under the same treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years
* Free and informed consent signed
* Histologically confirmed adenocarcinoma of the breast, metastatic or non-metastatic
* LVEF> 50% angioscintigraphy before the start of treatment with Herceptin ®,
* Overexpression of HER2 in the invasive component of the primary tumor (3 + 2 + according to ICH or with confirmation of positivity by FISH or CISH)
* Patient receiving treatment with Herceptin ®,
* Inclusion in the control group: patients treated with Herceptin ® episode without LV dysfunction,
* For the inclusion in the Group LV dysfunction: the appearance of a decrease in LVEF during treatment with Herceptin ®, angioscintigraphy identified.

Exclusion Criteria:

* Heart disease or serious medical conditions do not allow to administer Herceptin ® (documented history of heart failure, angina requiring treatment, severe dyspnoea at rest or oxygen dependency),
* History of ischemic heart disease or myocarditis
* Known allergy to trastuzumab, murine proteins or any of the excipients
* Patients with an indication against the MRI (claustrophobia, ferromagnetic foreign body, pacemaker or implantable defibrillator, known allergy to gadolinium salts)
* Renal impairment (creatinine clearance <60 ml / min according to the MDRD formula)
* Arrhythmia atrial fibrillation,
* Contraindications to the administration of Dotarem ®,
* Patient unable to give informed consent,
* Adult Trust,
* Pregnant or lactating
* Patient unable to undergo a medical for geographical, social or psychological.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Proportions of late enhancement in patients with LV dysfunction as Herceptin ® and in a control group consisting of patients who did not have LV dysfunction after 6 months under the same treatment. | 2 years
  A cardiac MRI is considered positive if demonstrated a late hyperintense from 15 to 20 minutes after injection of gadolinium chelate, whatever its size, topography subepicardial (intramyocardial) and without vascular systematization.
  The primary endpoint is the proportion of delayed enhancement in the LV dysfunction group and the control group.

SECONDARY OUTCOMES:
Proportion of patients recovering at 6 months in the absence of late enhancement signal in MRI heart after injection of gadolinium and compare the results of biological assays | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MANRIQUE Alain, Pr, Study Chair — GIP Cyceron; SWITSERS Odile, Dr, Principal Investigator — Centre François Baclesse
Locations (4):
- France (4):
  - Centre François Baclesse, Caen
  - Centre Georges-François Leclerc, Dijon
  - Clinique du Bois, Lille
  - CHU de NANCY, Nancy